CLINICAL TRIAL: NCT05887830
Title: Effect of Nivolumab vs Placebo in Patients With Acute Myocardial Infarction: A Randomized Clinical Trial
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YAN2023-0193
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Acute Anterior ST Segment Elevation Myocardial Infarction
Keywords: Nivolumab; acute anterior ST segment elevation myocardial infarction
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional drug treatment group (Experimental): The participants receive Nivolumab treatment. The active drug Nivolumab will be administered at a standard dose (5mg/kg) dissolved in 100ml 0.9%NaCl solution. Nivolumab was given at a rate of 15-25 drops per minute, and the intravenous infusion time exceeded 1 hour.
  Interventions: Drug: Nivolumab
- Placebo treatment group (Placebo Comparator): The participants receive placebo treatment. Patients assigned to the placebo treatment group will receive an intravenous infusion of 100 ml 0.9% NaCl solution at a rate of 15-25 drops/min for an IV infusion duration of more than 1 hour.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nivolumab — Single administration of Nivolumab on the third day of revascularization after acute anterior ST segment elevation myocardial infarction. The active drug Nivolumab will be administered at a standard dose (5mg/kg) dissolved in 100ml 0.9%NaCl solution. Nivolumab was given at a rate of 15-25 drops per minute, and the intravenous infusion time exceeded 1 hour.
  Arms: Interventional drug treatment group
Other: Placebo — Single administration of Placebo on the third day of revascularization after acute anterior ST segment elevation myocardial infarction. Patients assigned to the placebo treatment group will receive an intravenous infusion of 100 ml 0.9% NaCl solution at a rate of 15-25 drops/min for an IV infusion duration of more than 1 hour.
  Arms: Placebo treatment group

SUMMARY:
Myocardial infarction (MI) is a major contributor to morbidity and mortality in China. The goal of this interventional, randomised controlled clinical trial is to evaluate the effectiveness and safety of a single administration of Nivolumab to the patients presenting with an acute anterior ST-segmental elevated myocardial infarction. Researchers will investigate if Nivolumab treatment can effectively and safely reduce infarct size as well as improve cardiac function of the patients with acute myocardial infarction.

DETAILED DESCRIPTION:
The efficacy and safety of nivolumab as compared with placebo in the treatment of acute anterior ST segment elevation myocardial infarction are not known. In this phase 1/2, randomized, placebo-controlled, open-label trial, we randomly assigned adults with acute anterior ST segment elevation myocardial infarction to receive either nivolumab (5mg/kg for single administration) or placebo. The primary end points were difference in infarct size/LV mass% from baseline to 3 months after Nivolumab administration and the incidence of adverse events during 3 months after Nivolumab administration. Secondary end points included difference in LVEF%, LVESV/Body surface area, LVEDV/Body surface area, Trponin T and proBNP from baseline to 3 months after Nivolumab administration.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years;
2. Signed informed consent and expected compliance with protocol;
3. Acute anterior ST segment elevation myocardial infarction;
4. Emergency coronary angiography for revascularization of occlusive vessels within 24 hours of chest pain onset;
5. Left ventricular ejection fraction is less than 45% (LVEF≤45%) as revealed by Echo within 72 hours after revascularization.

Exclusion Criteria:

1. Cardiogenic shock;
2. Cardiac arrest/ventricular fibrillation;
3. History of severe renal failure, glomerular filtration rate (eGFR) < 30ml/min;
4. History of severe infection, hepatobiliary obstruction or malignant tumor;
5. Receiving immunosuppressive therapy;
6. Women who are pregnant or may become pregnant;
7. There are contraindications to study drugs or magnetic resonance examination;
8. No written informed consent was obtained.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
∆Infarct size/Left Ventricular mass% | 3 months
  Difference in Infarct size/Left ventricular mass% from baseline to 3 months after Nivolumab administration.
The incidence of adverse events | up to 3 months
  The incidence of adverse events during 3 months after Nivolumab treatment.

SECONDARY OUTCOMES:
∆Left ventricle ejection fraction% | 3 months
  Difference in Left ventricle ejection fraction% from baseline to 3 months after Nivolumab administration.
∆Left ventricle end systolic volume/Body surface area | 3 months
  Difference in Left ventricle end systolic volume/Body surface area from baseline to 3 months after Nivolumab administration.
∆Left ventricle end diastolic volume/Body surface area | 3 months
  Difference in Left ventricle end diastolic volume/Body surface area from baseline to 3 months after Nivolumab administration.
∆Troponin T | 3 months
  Difference in concentration of Troponin T from baseline to 3 months after Nivolumab administration.
∆proBNP | 3 months
  Difference in concentration of proBNP from baseline to 3 months after Nivolumab administration.

CONTACTS AND LOCATIONS:
Overall Officials: Xinyang Hu, PhD, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China

IPD SHARING:
Plan to Share IPD: No